CLINICAL TRIAL: NCT00137579
Title: Phase IV, Simple Blind, 2-Parallel Groups Randomized Trial to Evaluate the Safety and Effectiveness of the Intramuscular Vs Subcutaneous Route for the Administration of the Anti-Flu Vaccine in Patients Receiving Oral Anticoagulation
Brief Title: Safety of the Intramuscular Route of the Anti-Flu Vaccine in Patients Receiving Oral Anticoagulation Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catalan Institute of Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SINGRIP03
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2003-01

CONDITIONS: Influenza
Keywords: Influenza Vaccines; Acenocoumarol; Drug Administration Routes; Anticoagulants
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Procedure: Influenza vaccine intramuscular administration route

SUMMARY:
Until now, the best administration route of the anti-flu vaccine for patients receiving long term oral anticoagulation therapy has been the subcutaneous one; the intramuscular route has not been recommended because it may increase the risk of muscular haematoma. Although this practice is widely extended, no significant differences between the safety of both routes have been found. Some authors, analysing a small group of patients, affirm that the anti-flu vaccine can be administered safely by the intramuscular route on patients receiving long term oral anticoagulation therapy, while a previous opinion article recommended the subcutaneous route without any scientific evidence. Due to this, the investigators have done a clinical trial with the aim of determining the safety and effectiveness of the flu-vaccine intramuscular route in patients receiving long term oral anticoagulation therapy and also to analyse the possible interactions between the vaccine and the oral anticoagulant treatment.

DETAILED DESCRIPTION:
Phase IV, simple blind, 2-parallel groups, multicentric randomized trial where each patient will receive a single dose of the recommended by the WHO anti-flu vaccine for the 2003-2004 period, the control group will receive it subcutaneous and intervention group intramuscular. The assignation to each group will be randomized. The study included 4 basic areas of Barcelona city. Three visits have been scheduled for each patient: moment 0, 24 hours and 10 days after the vaccination, and a 7 month follow up period to control the incidence of the flu.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral anticoagulation therapy
* Patients who agree to be vaccinated
* Patients who agree to participate in the study
* Patients older than 18

Exclusion Criteria:

* Allergy or hypersensibility to egg, chicken proteins, any component of the vaccine (neomycin, octoxinol-9 or formaldehyd)
* INR greater than 4 in the past 2 months
* Previous major bleeding
* Patients with dementia or with legal tutoring

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216
Dates: Start 2003-09; Study Completion 2004-05

PRIMARY OUTCOMES:
local pain (scores greater than 3 in the analogic visual scale of pain)
microbiologically diagnosed flu (yes/no)
International Normalized Ratio (INR) to check the interaction between the vaccine and the oral anticoagulation therapy

SECONDARY OUTCOMES:
increase of the arm perimeter greater than 1 cm
local elemental skin lesions

CONTACTS AND LOCATIONS:
Overall Officials: Josep Casajuana, Physician, Principal Investigator — Catalan Institute of Health; Elvira Givert, Nurse, Study Chair — Catalan Institute of Health; Josep Franch, Physician, Study Chair — Catalan Institute of Health; Clara Sala, Nurse, Study Chair — Catalan Institute of Health; Miriam Aballi, Physician, Study Chair — Catalan Institute of Health; Begoña Iglesias, Physician, Study Chair — Catalan Institute of Health; Joan Antoni Valles, Physician, Study Chair — Catalan Institute of Health; Maria del Mar Piqueras, Physician, Study Chair — Catalan Institute of Health; Paz Escobar, Nurse, Study Chair — Catalan Institute of Health; Antonia Moreno, Nurse, Study Chair — Catalan Institute of Health; Montserrat Català, Nurse, Study Chair — Catalan Institute of Health; Anna Maria Ramirez, Nurse, Study Chair — Catalan Institute of Health; Maria Queralt Capdevila, Nurse, Study Chair — Catalan Institute of Health; Merce Botinas, Physician, Study Chair — Catalan Institute of Health; Lilia Villagrassa, Nurse, Study Chair — Catalan Institute of Health; Josep Maria Segura, Physician, Study Chair — Catalan Institute of Health; Maria del Mar Ballester, Physician, Study Chair — Catalan Institute of Health; Gustavo Losada, Physician, Study Chair — Catalan Institute of Health; Maria Teresa Maudos, Physician, Study Chair — Catalan Institute of Health
Locations (4):
- Spain (4):
  - Raval Nord, Barcelona, Barcelona
  - Raval Sud, Barcelona, Barcelona
  - Gotic, Barcelona, Barcelona
  - Casc Antic, Barcelona, Barcelona

REFERENCES:
- [Derived] Casajuana J, Iglesias B, Fabregas M, Fina F, Valles JA, Aragones R, Benitez M, Zabaleta E. Safety of intramuscular influenza vaccine in patients receiving oral anticoagulation therapy: a single blinded multi-centre randomized controlled clinical trial. BMC Blood Disord. 2008 May 29;8:1. doi: 10.1186/1471-2326-8-1. PMID 18507871